CLINICAL TRIAL: NCT02151578
Title: Home and Community Management of Fevers/Malaria and Pneumonia in Children Under-five: a Cluster Randomised Controlled Trial of an Integrated Approach in a Rural District of Burkina Faso
Brief Title: Home Management of Malaria and Pneumonia
Acronym: HMM/P
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: World Health Organization (Other)
Responsible Party: Principal Investigator, Sodiomon B. Sirima, Dr, World Health Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMMP001; A70210 (Other: WHO-TDR)
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Malaria; Pneumonia
Keywords: Impact of home management of malaria and pneumonia on child mortality; home management of malaria and pneumonia
MeSH Terms: conditions — Malaria; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- nothing at home level (No Intervention): No intervention at community level. The study drugs (arthemeter/Lumefantrine and Cotrimoxazole) available at the health facility drug stores level and prescribed exclusively to sick children attending to the health facility for care seeking. No Community Heath Worker /Key Opinion leader (CHWs/KOLs) selected in those clusters
- Home management of malaria (Experimental): At the community level, the Community health workers/ keay opinion leader (HWs/KOLs) trained and equipped to provide the antimalarial drug (arthemeter/Lumefantrine ) to any child with fever ("hot body") without any other signs of complications like impaired consciousness, convulsions, etc
  Interventions: Other: home/community case management
- Home management of malaria and pneumonia (Experimental): At the community level, the Community health workers/ key opinion leader (HWs/KOLs) trained and equipped to provide the antimalarial drug (arthemeter/Lumefantrine ) or antibiotic (Cotrimoxazole) to any child with fever ("hot body") without any other signs of complications like impaired consciousness, convulsions, etc. The treatment decision making for the CHWs/KOLs based on the algorithm
  Interventions: Other: home/community case management

INTERVENTIONS:
Other: home/community case management
  Arms: Home management of malaria; Home management of malaria and pneumonia

SUMMARY:
A well-implemented community-based program of early and appropriate treatment of fevers/malaria episodes and pneumonia,will improve child survival as measured by a reduction of the less than five mortality rate.

DETAILED DESCRIPTION:
An integrated approach of home and community management of malaria and pneumonia may increase the proportion of children receiving prompt treatment; improve child survival as measured by a reduction of the under five mortality rate. To test this hypothesis, a cluster randomised controlled trial will be performed, involving children less than 5 years of age, in Burkina Faso using a community-based supplying community health workers (CHWs), a core group of mothers (KOLs) with Coartem and cotrimoxazole specially packed in age-specific blisters containing a full course of treatment. The study will be carried out in 111 clusters of a rural district in Burkina Faso where malaria and pneumonia are two major mortality causes in under five mortality.

ELIGIBILITY:
Inclusion Criteria:

* living in one of the study cluster (villages)
* no story of allergy to any of the study drugs
* history of fever or body temperature >= 38.5°C

Exclusion Criteria:

* signs of severity/complications like impaired consciousness, convulsions, fast breathing etc

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11500 (Actual)
Dates: Start 2009-01; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of death in children aged 6 to 59 months | 12 months
  annual crude mortality rate in children aged 0 to 6 months in the different study arms

SECONDARY OUTCOMES:
- specific mortality preceded by acute febrile illness of children aged 6 to 59 months - severe malaria cases at community level | 12 months

OTHER OUTCOMES:
Adverse events at community level consecutive to the administration of the cotrimoxazole and arthemeter/lumefantrine | 7 days after the administration of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Sodiomon Bienvenu SIRIMA, MD, PhD, Principal Investigator — Groupe de Recherche Action en santé (GRAS), 06 BP 10248 Ouagadougou 06, Burkina Faso
Locations (1):
- Groupe de Recherche Action en Sante (GRAS sarl), Ouagadougou, Kadiogo, Burkina Faso

REFERENCES:
- [Derived] Oliphant NP, Manda S, Daniels K, Odendaal WA, Besada D, Kinney M, White Johansson E, Doherty T. Integrated community case management of childhood illness in low- and middle-income countries. Cochrane Database Syst Rev. 2021 Feb 10;2(2):CD012882. doi: 10.1002/14651858.CD012882.pub2. PMID 33565123